CLINICAL TRIAL: NCT03848156
Title: In Depth Characterisation of Nasal Polyps in Patients With and Without Aspirin-exacerbated Respiratory Disease - a Pilot Study
Brief Title: Characterisation of Nasal Polyps in Patients With and Without Aspirin-exacerbated Respiratory Disease
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Sven Schneider, MD, Principal Investigator, Medical University of Vienna
Other Study IDs: AERD2019
Record Dates: First submitted 2019-02-13; First posted 2019-02-20 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Polyp Sinus
MeSH Terms: interventions — Biopsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Polyp biopsy, blood, nasal secretion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- CRSwNP AERD allergic: Patients suffering from chronic rhinosinusitis with nasal polyps, allergy and aspirin exacerbated respiratory disease - biopsy for RNA sequencing
  Interventions: Other: biopsy
- CRSwNP AERD non-allergic: Patients suffering from chronic rhinosinusitis with nasal polyps without allergy and aspirin exacerbated respiratory disease - biopsy for RNA sequencing
  Interventions: Other: biopsy
- CRSwNP non-allergic: Patients suffering from chronic rhinosinusitis with nasal polyps without allergy - biopsy for RNA sequencing
  Interventions: Other: biopsy
- CRSwNP allergic: Patients suffering from chronic rhinosinusitis with nasal polyps with allergy - biopsy for RNA sequencing
  Interventions: Other: biopsy

INTERVENTIONS:
Other: biopsy — Biopsy of nasal polyp for RNA sequencing

SUMMARY:
Prevalence of aspirin-exacerbated respiratory disease (AERD) is 16% amongst patients suffering from chronic rhinosinusitis with nasal polyps (CRSwNP). The mechanisms underlying the observed dysregulation of pro and anti-inflammatory pathways in AERD are still not fully understood. To address this and also to identify potential factors characterizing the disease the investigators plan to prospectively collect blood samples, nasal secretions as well as nasal biopsies from allergic, non-allergic and AERD patients suffering from CRSwNP. Initially, polyps of aforementioned patients will be subjected to RNA sequencing analysis using microarray technology. Once distinct factors are identified in nasal polyp tissue, their presence will be assessed in nasal secretions and serum of the respective patients to investigate their potential role as biomarkers. Furthermore presence of these parameters will be confirmed in situ in biopsies by confocal microscopy. Knowledge about factors differently upregulated in polyp tissue from AERD may contribute to a better understanding of the underlying mechanism of the disease.

DETAILED DESCRIPTION:
Chronic rhinosinusitis (CRS) with (w) and without (s) nasal polyps (NP) in its different shapes is currently affecting up to 16% of the total population of the United States and around 11% of the population in Europe. However CRS may also be associated with hypersensitivity to aspirin and other non-selective cyclooxygenase inhibitors. This syndrome of combined CRSwNP, asthma and intolerance to inhibitors of the cyclooxygenase-1 enzyme was termed Samter's triad or aspirin-exacerbated respiratory disease (AERD). AERD is thought to affect around 16% of patients suffering from CRSwNP, around 7% of adult asthmatic patients and 0.3-2.5% of the general population. One characteristic feature of this disease is the presence of nasal polyps that frequently relapse after surgery rendering this disease difficult to manage. Despite its relatively high prevalence, the pathophysiologic mechanisms are yet not fully understood. In this respect, an overproduction of and overresponsiveness to cysteinyl leukotrienes accompanied by and underproduction of and underresponsiveness to prostaglandins was observed in AERD patients.This indicates a dysregulation of pro and anti-inflammatory pathways. However the mechanism and the cells involved in causing this imbalance are still not clear.

The availability of gene-chip microarray technology allows for quantitatively and simultaneously monitoring of the expression of thousands of genes and has greatly contributed to the understanding of pathological mechanisms. In this context, analysis of nasal polyps from allergic patients has shown that genes involved in deregulated cell growth similar to neoplastic growth are upregulated in this tissue. Furthermore very recently, profiling of CRS samples by single-cell RNA sequencing revealed a significant loss of epithelial ecological diversity in nasal polyps. The authors suggest that basal cells form memories of chronic exposure to an inflammatory environment and shift the cellular ecosystem towards propagating the disease. However polyps from AERD patients which show a different clinical and most likely also pathophysiological profile have not been included in this study. Given the prevalence of 15% amongst CRSwNP patients and the impaired quality of life of AERD patients it would be desirable to understand the difference between AERD and CRSwNP without AERD at a molecular level and also to potentially find biomarkers that uniquely identify patients suffering from AERD disease.

Therefore, the investigators plan to prospectively collect blood samples, nasal secretions as well as nasal biopsies from allergic, non-allergic and AERD patients suffering from CRSwNP. Initially, RNA sequencing will be performed using microarray technology in biopsies of those patients. Once parameters are identified, the investigators will investigate if a similar pattern can also be detected in nasal secretions and/or serum of the respective patients to investigate their potential as biomarkers. Furthermore presence of these parameters will be confirmed in situ in biopsies by confocal microscopy.

ELIGIBILITY:
Inclusion criteria:

* Male or Female
* Age: 18-90
* Willingness to participate in the study
* Suffering from CRSwNP (with or without prior history of surgery for nasal polyposis)
* Allergic or non-allergic: if no recent allergy test is available (max. two years old) the presence or absence of allergy will be determined by skin prick test and by ImmunoCAP for allergen-specific serum immunoglobulin E (IgE) levels in addition to assessment of patients's history by questionnaire.
* Suffering from AERD or not as confirmed by provocation testing

Exclusion criteria:

* Children
* Pregnant women - the presence of a known pregnancy will be assessed during the visit by questionnaire
* A mental condition rendering the subject unable to understand the nature, scope and possible consequences of the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients suffering from chronic rhinosinusitis with nasal polyps with/without AERD and with/without allergy
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
RNA Sequencing of polyps using Illumina platform | patients will be recruited over the course of one year until 20 patients have been reached. Each patient will be sequenced when the sample is received.
  Differences in expression patterns in RNA expression in the 4 groups assessed using Illumina platform for RNA sequencing

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided